CLINICAL TRIAL: NCT01232283
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Evaluate Safety and Effectiveness of Oral Apremilast (CC-10004) in Patients With Moderate to Severe Plaque Psoriasis.
Acronym: ESTEEM 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-009
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2020-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apremilast (Experimental): Participants were initially randomized 2:1 and received apremilast 30 mg twice a day (BID). Participants maintained dosing through Week 32. At Week 32, responders, those with a Psoriasis Area Severity Index response -≥75 (PASI-75) and partial responders (≥PASI-50) were re-randomized 1:1 to apremilast 30 mg BID or matching placebo (treatment withdrawal). Participants could resume apremilast 30 mg BID at the time of loss of 50% of improvement in PASI score response which was observed at Week 32 compared to baseline), and no later than Week 52. At Week 52, the non-responders (<PASI-50) had the option of adding topical therapies and/or phototherapy to their treatment regimen. Those re-randomized to apremilast 30 mg BID continued dosing through Week 52. At Week 52, participants continued treatment with apremilast 30 mg BID.
  Interventions: Drug: Apremilast; Drug: Placebo; Other: Topical or Phototherapy Therapy
- Placebo (Placebo Comparator): Participants will be initially randomized to placebo, identically matching during Weeks 0-16. At Week 16, Placebo participants will be switched to receive apremilast 30 mg BID. All participants will maintain Apremilast dosing through Week 32. At Week 32, participants originally randomized to placebo at baseline (Week 0) and are considered non-responders i( < PASI-50) will have the option of adding topical therapies and/or phototherapy to their Apremilast treatment regimen. At Week 52, all participants will continue treatment with apremilast 30 mg BID. Participants will be followed and evaluated for safety and efficacy for up to an additional 4 years (years 2 through 5).
  Interventions: Drug: Apremilast; Drug: Placebo; Other: Topical or Phototherapy Therapy

INTERVENTIONS:
Drug: Apremilast — Apremilast 30mg by mouth (PO) twice a day (BID) for 32 weeks
  Other Names: CC-10004; Otezla
Drug: Placebo — Identically matching placebo by mouth BID for first 16 weeks. Placebo participants will be switched to receive apremilast 30 mg BID at Week 16-32.
Other: Topical or Phototherapy Therapy — Topical therapies such as low-potency or weak corticosteroids or phototherapies such as light therapy are added for non-responders at Week 32, (< PASI-50) and added to their treatment regimen. The decision to add these treatments during this phase can only be made at the Week 32 visit.

SUMMARY:
This study will evaluate the effects of an experimental (being tested) study drug called apremilast. Apremilast works by lowering some of the chemicals that affect psoriasis and therefore improves the symptoms of psoriasis. The purpose of this study is to test apremilast and compare its effects to placebo (an inactive substance which contains no medicine but is in the same form as the drug). This study will test efficacy (improvement of signs and symptoms) and safety of apremilast in patients with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 years of age at the time of signing the informed consent document
2. Diagnosis of chronic plaque psoriasis for at least 12 months prior to Screening

   a. Have moderate to severe plaque psoriasis at Screening and Baseline
3. Must meet all laboratory criteria
4. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use 2 forms of contraception as described by the Study Doctor while on study medication and for at least 28 days after taking the last dose of study medication
5. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex condom or any nonlatex condom NOT made out of natural [animal] membrane [eg, polyurethane]) while on study medication and for a least 28 days after the last dose of study medication.

Exclusion Criteria:

1. Other than psoriasis, history of any clinically significant (as determined by the Investigator) or other major uncontrolled disease.
2. Pregnant or breast feeding
3. History of allergy to any component of the study drug
4. Hepatitis B surface antigen positive at Screening
5. Anti-hepatitis C antibody positive at Screening
6. Active tuberculosis (TB) or a history of incompletely treated TB
7. Clinically significant abnormality on 12-Lead ECG at Screening
8. Clinically significant abnormal chest x-ray
9. History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency
10. Active substance abuse or a history of substance abuse within 6 months prior to Screening
11. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening
12. Malignancy or history of malignancy (except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and treated [ie, cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years)
13. Psoriasis flare or rebound within 4 weeks prior to Screening
14. Evidence of skin conditions that would interfere with clinical assessments
15. Topical therapy within 2 weeks of randomization
16. Systemic therapy for psoriasis within 4 weeks prior to randomization
17. Use of phototherapy within 4 weeks prior to randomization (ie, UVB, PUVA)
18. Adalimumab, etanercept, infliximab, or certolizumab pegol within 12 weeks prior to randomization
19. Alefacept, briakinumab, or ustekinumab within 24 weeks prior to randomization
20. Use of any investigational drug within 4 weeks prior to randomization
21. Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources
22. Prior treatment with apremilast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2012-03-15 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (46):
- United States (19):
  - Arizona Skin and Laser Therapy Inst., Ltd., Phoenix, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Florida Academic Dermatology Center, Miami, Florida
  - Advanced Medical Research, Atlanta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Northwestern University Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - Austin Dermatology Associates, Austin, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Medical Research, Norfolk, Virginia
- Medizinische Universitat Wien, Universitatsklinik fur Dermatologie. Abteilung fur Immundermatologie, Vienna, Austria
- Canada (7):
  - Northwest Dermatology and Laser Centre, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - NewLab Clinical Research, St. John's, Newfoundland and Labrador
  - Skin Center for Dermatology, Peterborough, Ontario
  - Windsor Clinical Research Inc., Winsor, Ontario
  - Q & T Research Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain CRDQ, Québec
- Bispebjerg Hospital, Copenhagen, Denmark
- France (3):
  - Centre d'lnvestigation Clinique, Hopital Jean Minjoz, Besançon
  - Hospital haut leveque, Pessac
  - Larrey University Hospital, Toulouse
- Germany (5):
  - Dr. med. Beatrice Gerlach, Dresden
  - Universitatsklinikum Hamburg-Eppendorf / IVDP, Hamburg
  - Universitäts-Hautklinik Kiel, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Hautarztpraxis Mahlow, Mahlow
- Italy (3):
  - Universita degli Studi di Napoli Federico II, Napoli
  - Istituto Dermatologico San Gallicano IRCCS Dermatologia Clinica, Rome
  - A.O.U. Integrata di Verona Universitá degli Studi di Verona Sezione di Dermatologia e Venerologia, Verona
- Spain (5):
  - Hospital Abente y Lago, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Universitari Germans Trias i Pujol, Badalona (Barcelona)
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - Hopitaux Universitaires de Geneve-HUG, Geneva
  - University of Zurich Hospital, Zurich

REFERENCES:
- [Background] Reich K, Mrowietz U, Menter A, Griffiths CEM, Bagel J, Strober B, Nunez Gomez N, Shi R, Guerette B, Lebwohl M. Effect of baseline disease severity on achievement of treatment target with apremilast: results from a pooled analysis. J Eur Acad Dermatol Venereol. 2021 Dec;35(12):2409-2414. doi: 10.1111/jdv.17520. Epub 2021 Aug 23. PMID 34255891
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 46 study centers in 9 countries.
Pre-assignment Details: Participants were eligible who had moderate to severe plaque psoriasis.
Groups:
- Apremilast: Participants initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
- Placebo: Participants initially randomized to identically matching placebo tablets (PBO) BID during the Placebo controlled Phase (Weeks 0-16)
- Apremilast-Apremilast: Participants who were initially randomized to apremilast 30 mg tablets BID during the Placebo-controlled Phase (Weeks 0-16) remained on apremilast 30 mg BID during the Maintenance Phase (Weeks 16-32).
- Placebo-Apremilast: Participants who were initially randomized to placebo BID during the Placebo-controlled Phase (Weeks 0-16) were switched after 16 weeks of treatment to apremilast 30 mg BID and continued dosing with apremilast 30 mg BID during the Maintenance Phase (Weeks 16-32).
- APR-APR-Re-randomized to PBO: Participants who were initially randomized to apremilast 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with apremilast 30 mg BID through the Maintenance Phase (Weeks 16-32). At week 32, those participants who were considered responders (ie, having a ≥PASI-50 response) were re-randomized to placebo during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who lost their PASI-50 improvement achieved at Week 32, were switched back to apremilast 30 mg BID at the time the loss was observed. Those participants who did not lose their PASI-50 response remained on placebo until Week 52. All participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and received apremilast 30 mg BID for the remainder of their participation.
- APR-APR Re-randomized to APR: Participants who were initially randomized to apremilast 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with apremilast 30 mg BID through the Maintenance Phase (Weeks 16-32). At week 32, those participants who were considered responders (ie, having a ≥PASI-50 response) were re-randomized to apremilast during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and continued on apremilast 30 mg BID for the remainder of their participation.
- APR-APR-APR + Optional Topicals/Phototherapy: Participants who were initially randomized to apremilast 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with apremilast 30 mg BID through the Maintenance Phase (Weeks 16-32). At Week 32, those participants who were considered non-responders (ie, having a response of <PASI-50), remained on apremilast 30 mg BID and were given the option of adding topical therapies and/or phototherapy to their regimen. Those participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and continued on apremilast 30 mg BID for the remainder of their participation.
- PBO-APR-APR + Optional Topicals/Phototherapy: Participants who were initially randomized to placebo BID during the 16-week Placebo-controlled Phase (Weeks 0-16) were switched after 16 weeks of treatment to apremilast 30 mg BID and continued dosing with apremilast 30 mg BID during the Maintenance Phase (Weeks 16-32). At week 32, all participants were to maintain apremilast 30 mg BID; those who were non-responders (having a response of <PASI-50), remained on apremilast 30 mg BID and were given the option of adding topical therapies and/or phototherapy to their regimen. A subset of these non-responders received additional topicals or phototherapy. All participants who completed the Randomized Withdrawal Phase at week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and continued on apremilast 30 mg BID for the remainder of their participation
- Apremilast (Long-Term Extension Phase): Participants who were initially randomized to APR 30 mg BID during the 16-week placebo-controlled phase (Weeks 0-16) continued receiving APR 30 mg BID through the Maintenance Phase (weeks 16-32) and apremilast 30 mg tablets or placebo during the Randomized Withdrawal Phase were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and remained on APR 30 mg BID for the remainder of their participation.
- Placebo-Apremilast (Long-term Extension): Participants who were initially randomized to identically matching placebo BID during the Placebo-controlled Phase (Weeks 0-16) were switched at Week 16 to apremilast 30 mg BID during the Maintenance Phase, received apremilast 30 mg PO BID during the Randomized Withdrawal Phase and then received apremilast 30 mg tablets BID in the long-term extension phase from weeks 52-260.
Period: Placebo Controlled Phase (Weeks 0-16)
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR Re-randomized to APR | APR-APR-APR + Optional Topicals/Phototherapy | PBO-APR-APR + Optional Topicals/Phototherapy | Apremilast (Long-Term Extension Phase) | Placebo-Apremilast (Long-term Extension)
Started | 275 | 138 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Apremilast | 272 (1 protocol violation occurred) | 136 (1 protocol violation occurred) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 239 | 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 36 | 26 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 12 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance with study drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Phase (Weeks16-32)
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR Re-randomized to APR | APR-APR-APR + Optional Topicals/Phototherapy | PBO-APR-APR + Optional Topicals/Phototherapy | Apremilast (Long-Term Extension Phase) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 234 (5 participants discontinued after Week 16 but prior to entry into the Maintenance Phase) | 108 (4 participants discontinued after Week 16 but prior to entry into the Maintenance Phase) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 194 | 100 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 40 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 19 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal Phase(Weeks 32-52)
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR Re-randomized to APR | APR-APR-APR + Optional Topicals/Phototherapy | PBO-APR-APR + Optional Topicals/Phototherapy | Apremilast (Long-Term Extension Phase) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 0 | 0 | 62 (4 participants discontinued after Week 32 but prior to entry into the Randomized Withdrawal Phase) | 61 (13 participants discontinued after Week 32 but prior to entry into the Randomized Withdrawal Phase) | 58 | 96 | 0 | 0
Treated With APR+ Topicals/Phototherapy | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 17 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 50 | 56 | 41 | 84 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 5 | 17 | 12 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 4 | 0 | 13 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 4 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Long-Term Extension Phase (Weeks 52-260)
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR Re-randomized to APR | APR-APR-APR + Optional Topicals/Phototherapy | PBO-APR-APR + Optional Topicals/Phototherapy | Apremilast (Long-Term Extension Phase) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 137 | 80
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 | 61
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 30
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were randomized as specified in the protocol. Those who were randomized in error and did not receive any dose of Investigational product (IP) were excluded from FAS. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS.
Groups:
- Apremilast: Participants were initially randomized to Apremilast (APR) 30 mg tablets BID during the Placebo-controlled Phase (weeks 0-16)
- Placebo: Participants were initially randomized to placebo tablets BID during the Placebo controlled Phase (weeks 0-16).
- Total: Total of all reporting groups
Arm/Group | Apremilast | Placebo | Total
Number analyzed (Participants) | 274 | 137 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.05) | 45.7 (13.38) | 45.4 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 37 | 135
  Male | 176 | 100 | 276
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 8 | 6 | 14
  Black or African American | 13 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 250 | 128 | 378
  Other-not specified | 1 | 0 | 1
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] — All participants enrolled were required to have a diagnosis of plaque psoriasis at least 12 months prior to screening, but the duration was not required for enrollment. Overall baseline population for duration of plaque psoriasis in the apremilast arm were 271 participants and 135 for those in the placebo arm.
  years | 17.94 (11.367) | 18.68 (12.088) | 18.19 (11.602)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least a 75% Improvement (Response) in the Psoriasis Area Severity Index (PASI-75) at Week 16 From Baseline
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at week 16. The improvement in PASI score was used as a measure of efficacy. The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement is missing.
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward (LOCF) imputation was used. .
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 274 | 137
percentage of participants | 28.8 | 5.8
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 23.0, 95% CI 2-sided [16.3 to 29.6]

2. Secondary Outcome: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) With at Least 2 Points Reduction From Baseline
Description: The sPGA was a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. When making the assessment of overall severity, the Investigator must have factored in areas that have already been cleared (ie, have scores of 0) and not just evaluate remaining lesions for severity, ie, the severity of each sign was averaged across all areas of involvement, including cleared lesions. In the event of different severities across disease signs, the sign that is the predominant feature of the disease should be used to help determine the sPGA score.
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants were initially randomized to identically matching PBO tablets twice daily BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 274 | 137
percentage of participants | 20.4 | 4.4
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 16.1, 95% CI 2-sided [10.2 to 21.9]

3. Secondary Outcome: Percent Change From Baseline in the Affected Body Surface Area (BSA) at Week 16
Description: BSA was a measurement of involved skin. The overall BSA affected by psoriasis was estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area.
  BSA percent change from baseline (Visit 2 Week 0) was determined at each visit of the study, which is calculated as 100*(visit BSA - baseline BSA) / baseline BSA (%).
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Participants with a baseline value and at least 1 postbaseline value were included. Last observation carried forward imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Participants were initially randomized to placebo (PBO) tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 269 | 136
percent change | -48.40 (2.636) | -6.25 (3.710)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The model included treatment group as a factor and the baseline value as a covariate. The estimation and p-value were adjusted by the covariate; Difference in LS Mean = -42.15, 95% CI 2-sided [-51.11 to -33.20]

4. Secondary Outcome: Percent Change From Baseline in the Psoriasis Area Severity Index (PASI) Score at Week 16
Description: Psoriasis Area Severity Index (PASI) scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score. The PASI score was set to missing if any severity score or degree of involvement is missing.
Time Frame: Baseline and Week 16
Population: FAS consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward (LOCF) imputation was used. Participants with a baseline value and at least 1 postbaseline value are included.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Participants were initially randomized to placebo tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 269 | 136
percent change | -50.8 (2.23) | -16.0 (3.15)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -34.8, 95% CI 2-sided [-42.4 to -27.2]

5. Secondary Outcome: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score (PASI-50) at Week 16 From Baseline
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement is missing.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Groups:
- Apremilast: Participants were initially randomized to apremilast 30 mg tablets BID during the Placebo-controlled Phase (Weeks 0-16)
- Placebo: Participants were initially randomized to identically matching placebo tablets BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 274 | 137
Percentage of Participants | 55.5 | 19.7
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 35.8, 95% CI 2-sided [26.9 to 44.7]

6. Secondary Outcome: Change From Baseline in Pruritus Visual Analog Scale (VAS) Score at Week 16
Description: The Pruritus Visual Analog Scores (VAS) were used to measure the amount of itching and discomfort a participant experiences. Participant's Assessment of Pruritus (Itch) asked: On average, how much itch have you had because of your condition in the past week? All VAS values range from 0 to 100. Higher scores correspond to more severe symptom or disease. Change from baseline was calculated for the VAS scale, where change = visit value - baseline value.
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward imputation was used. Participants with a baseline value and at least 1 postbaseline value are included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants were initially randomized to identically matching PBO tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 268 | 133
units on a scale | -33.5 (2.08) | -12.2 (2.95)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -21.3, 95% CI 2-sided [-28.4 to -14.2]

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the subject is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 267 | 131
units on a scale | -6.7 (0.37) | -2.7 (0.53)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -4.0, 95% CI 2-sided [-5.3 to -2.8]

8. Secondary Outcome: Change From Baseline in the Mental Component Summary (MSC) Score of the Medical Outcome Study Short Form 36-item (SF-36) Health Survey Version 2.0 at Week 16
Description: The SF-36 was a 36-item general health instrument and consists of 8 scales: physical function (PF), role limitations-physical (RP), vitality (VT), general health perceptions (GH), bodily pain (BP), social function (SF), role limitations-emotional (RE), and mental health (MH). Scale scores range from 0 to 100, with higher scores indicating better health. Two overall summary scores were obtained - a Physical Component Summary score (PCS) and a Mental Component Summary score (MCS).
  Scores from the 8 scales, PCS and MCS were transformed to the norm-based scores using weights from U.S. general population, with 50 as the average and 10 as the standard deviation, higher scores indicating better health. For norm based scores, change from baseline were calculated for the 8 scales and the two summary scales, where change = visit value - baseline value.
Time Frame: Baseline to Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Apremilast: Participants were initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 267 | 131
units on a scale | 2.60 (0.563) | -0.03 (0.804)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p = 0.0078, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = 2.63, 95% CI 2-sided [0.69 to 4.56]

9. Secondary Outcome: Percentage of Participants Who Achieved Both a 75% Improvement (Response) in the PASI and sPGA Score of Clear (0) or Almost Clear (1) With at Least 2 Points Reduction at Week 16 From Baseline
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. See Outcome measure #1 for further description.
  sPGA is a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. See Outcome Measure #2 for further description.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 274 | 137
percentage of participants | 18.6 | 4.4
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 14.2, 95% CI 2-sided [8.5 to 20.0]

10. Secondary Outcome: Time to Loss of Effect (Loss of 50% Improvement in PASI Score Obtained at Week 32 Compared to Baseline) During the Randomized Treatment Withdrawal Phase
Description: Time to loss was the time between the re-randomization date and the date of the first assessment with loss of 50% PASI improvement (event), or the time between the re-randomization date and the date of the last PASI assessment in the randomized withdrawal phase prior to addition of topical/phototherapy or other effective psoriasis therapies, or resumption of apremilast 30 mg BID, or discontinuation, or Week 52 if no loss (censored), whichever was earlier
Time Frame: Weeks 32 to Week 52
Population: Analysis population consisted of participants who were re-randomized to placebo or Apremilast 30mg BID at Week 32.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- APR-APR Re-randomized to PBO: Participants who were initially randomized to apremilast 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with apremilast 30 mg BID through the Maintenance Phase (Weeks 16-32). At week 32, those participants who were considered responders (ie, having a ≥PASI-50 response) were re-randomized to placebo during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who lost their PASI-50 improvement achieved at Week 32, were switched back to apremilast 30 mg BID at the time the loss was observed. Those participants who did not lose their PASI-50 response remained on placebo until Week 52. All participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and received apremilast 30 mg BID for the remainder of their participation.
- APR-APR-Re-randomized to APR: Participants who were initially randomized to apremilast 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with apremilast 30 mg BID through the Maintenance Phase (Weeks 16-32). At week 32, those participants who were considered responders (ie, having a ≥PASI-50 response) were re-randomized to apremilast during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and continued on apremilast 30 mg BID for the remainder of their participation.
Arm/Group | APR-APR Re-randomized to PBO | APR-APR-Re-randomized to APR
Number analyzed (Participants) | 62 | 61
Weeks | 12.4 [8.3 to 20.1] | 21.9 [NA to NA] — The confidence interval was not calculated because there was no sufficient information from data for the confidence interval estimate
Statistical Analysis 1: Comparison: APR-APR Re-randomized to PBO vs APR-APR-Re-randomized to APR; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 7.700, 95% CI 2-sided [3.408 to 17.399]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in the Placebo Controlled Phase
Description: An AE was any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Baseline to Week 16
Population: Safety population consisted of all participants who were randomized and received at least one dose of Investigational Product (IP)
Measure: Number; unit: participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 272 | 136
participants
  Any TEAE | 185 | 82
  Any drug related TEAE | 106 | 29
  Any Severe TEAE | 12 | 6
  Any Serious TEAE | 5 | 3
  Any TEAE leading to drug interruption | 16 | 4
  Any TEAE leading to drug withdrawal | 15 | 7

12. Secondary Outcome: Number of Participants With Psoriasis Flare or Rebound in the Placebo Controlled Phase
Description: Psoriasis flare was defined as a sudden intensification of psoriasis requiring medical intervention, or a diagnosis of new generalized erythrodermic, inflammatory, or pustular psoriasis. Rebound is defined as a severe and sudden worsening of disease that occurs after treatment has been discontinued. Note categories below. [1] Psoriasis adverse events (ie, preferred term as Guttate psoriasis, Psoriasis, Pustular psoriasis) started on or after the first dose date and on or before the last dose date within the phase. [2] Psoriasis adverse events (ie, preferred term as Guttate psoriasis, Psoriasis, Pustular psoriasis, Rebound psoriasis) started after the last dose date for participants who discontinued within the phase. [3] PASI >= 125% of baseline score at any visit after the last dose date for participants who discontinued within the phase and were not included in [1] and/or [2].
Time Frame: Week 0 to Week 16
Population: Safety population, included all participants who were randomized and received at least one dose of IP. Participants with a PASI ≥ 125% of Baseline score after last dose who did not have psoriasis rebound captured as a Treatment Emergent Adverse Event.
Measure: Number; unit: participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 272 | 136
participants
  Participants with any psoriasis flare | 3 | 7
  Participants with any psoriasis rebound | 1 | 0
  PASI ≥ 125% of Baseline score after last dose | 1 | 2

13. Secondary Outcome: Number of Participants With TEAEs During the Apremilast-Exposure Period Through Week 260
Description: The Apremilast-exposure Period started on the date of the first dose of apremilast (Week 0 for participants originally randomized to apremilast or Week 16 for participants originally randomized to placebo) to the last dose of apremilast. Adverse events that started after 28 days of initiating placebo and before resuming apremilast treatment in the Randomized Treatment Withdrawal Phase (Weeks 32 to 52) were excluded in the Apremilast-exposure phase. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Week 0 to Week 260; The mean duration of exposure was 100.66 weeks.
Population: Apremilast participants as treated, which includes all participants who were randomized to (at Week 0) or treated with (at Week 16) apremilast 30 mg BID, and received at least one dose of apremilast after randomization or Week 16.
Measure: Number; unit: participants
Groups:
- Apremilast: Participants who received apremilast 30 mg BID at any time during the study. Participants initially randomized to placebo or apremilast 30 mg tablets BID during the 16-week placebo-controlled phase (Weeks 0-16) continued to receive apremilast 30 mg BID through the maintenance phase; during the randomized withdrawal phase (Weeks 32-52) participants were again randomized to either apremilast 30 mg BID or placebo and were transitioned to apremilast 30 mg BID after loss of response or in the long-term extension phase from Weeks 52-260,
Arm/Group | Apremilast
Number analyzed (Participants) | 380
participants
  Any TEAE | 316
  Any Drug-Related TEAE | 165
  Any Severe TEAE | 58
  Any Serious TEAE | 44
  Any Serious Drug-Related TEAE | 8
  Any TEAE Leading to Drug Interruption | 56
  Any TEAE Leading to Drug Withdrawal | 45
  Any TEAE Leading to Death | 1

14. Secondary Outcome: Number of Participants With Psoriasis Flare or Rebound in the Apremilast-Exposure Period
Description: as for outcome 12
Time Frame: Week 0 to Week 260
Population: The apremilast subjects as treated population, which includes all participants who were randomized to (at Week 0) or treated with (at Week 16) apremilast 30 mg BID, and received at least one dose of apremilast after randomization or Week 16.
Measure: Number; unit: participants
Groups:
- Apremilast: Participants who received apremilast 30 mg BID at any time during the study.
Arm/Group | Apremilast
Number analyzed (Participants) | 272
participants
  Participants with any psoriasis flare | 25
  Participants with any psoriasis rebound | 11
  PASI ≥ 125% of Baseline score after last dose | 12

ADVERSE EVENTS:
Time Frame: AEs are reported at: 1. Weeks 0-16: PBO-controlled phase 2. Weeks 32-52 Randomized Withdrawal participants re-randomized to PBO at Week 32 3. Weeks 0-260 APR-exposure period for participants randomized or switched to APR at any time during the study
Description: During the PBO-controlled Phase (Weeks 0-16), the mean duration of treatment for those randomized to APR 30 BID or PBO at Week 0, was 14.0 and 14.6, respectively; for those re-randomized to PBO at Week 32, the mean duration of PBO was 11.6 weeks; during the APR-Exposure Period (Weeks 0-260), the mean duration of exposure to APR was 100.66 weeks
Groups:
- Placebo: Weeks 0-16 (PBO-Controlled Phase): Participants randomized to identically matching placebo tablets BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast: Weeks 0-16 (PBO-Controlled Phase): Participants randomized to apremilast 30 mg tablets BID during the Placebo-controlled Phase (Weeks 0-16)
- APR-APR-PBO: Weeks 32-52 (Randomized Withdrawal Phase): Participants re-randomized to placebo tablets BID at Week 32. Includes data from Week 32 up to Week 52 when participants received placebo treatment.
- Apremilast: Weeks 0-260 (APR- Exposure Period ): Participants who received apremilast 30 mg tablets BID, regardless of when the apremilast exposure started (at Week 0 or at Week 16), up until Week 260. Adverse events associated with apremilast 30 mg treatment up to Week 260 were included. AEs that started more than 28 days after placebo treatment and prior to resuming apremilast were excluded for participants who were re-randomized to Placebo at Week 32.
Arm/Group | Placebo: Weeks 0-16 (PBO-Controlled Phase) | Apremilast: Weeks 0-16 (PBO-Controlled Phase) | APR-APR-PBO: Weeks 32-52 (Randomized Withdrawal Phase) | Apremilast: Weeks 0-260 (APR- Exposure Period )
Serious Adverse Events (participants affected / at risk) | 3/136 | 5/272 | 2/62 | 44/380
Other Adverse Events (participants affected / at risk) | 38/136 | 128/272 | 17/62 | 234/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Weeks 0-16 (PBO-Controlled Phase) (N=136) | Apremilast: Weeks 0-16 (PBO-Controlled Phase) (N=272) | APR-APR-PBO: Weeks 32-52 (Randomized Withdrawal Phase) (N=62) | Apremilast: Weeks 0-260 (APR- Exposure Period ) (N=380)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Weeks 0-16 (PBO-Controlled Phase) (N=136) | Apremilast: Weeks 0-16 (PBO-Controlled Phase) (N=272) | APR-APR-PBO: Weeks 32-52 (Randomized Withdrawal Phase) (N=62) | Apremilast: Weeks 0-260 (APR- Exposure Period ) (N=380)
Diarrhoea (Gastrointestinal disorders) | 8 | 43 | 1 | 62
Nausea (Gastrointestinal disorders) | 9 | 50 | 2 | 68
Vomiting (Gastrointestinal disorders) | 5 | 14 | 0 | 27
Bronchitis (Infections and infestations) | 0 | 4 | 1 | 29
Nasopharyngitis (Infections and infestations) | 6 | 20 | 5 | 69
Upper respiratory tract infection (Infections and infestations) | 6 | 13 | 1 | 53
Urinary tract infection (Infections and infestations) | 0 | 5 | 1 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 1 | 19
Headache (Nervous system disorders) | 1 | 17 | 0 | 28
Tension headache (Nervous system disorders) | 2 | 20 | 0 | 31
Psoriasis (Skin and subcutaneous tissue disorders) | 7 | 3 | 1 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.